CLINICAL TRIAL: NCT00344734
Title: Effects of Acute L-NMMA Treatment on Renal Hemodynamics, Sodium and Water Excretion and Plasma Levels of Vasoactive Hormones in Patients With Congestive Heart Failure and Healthy Controls
Brief Title: Effects of Acute L-NMMA Treatment on Renal Hemodynamics and Vasoactive Hormones in Patients With Congestive Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MED.RES.HOS.1997.03.JNB
Record Dates: First submitted 2006-06-24; First posted 2006-06-27 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2006-06

CONDITIONS: Congestive Heart Failure
Keywords: Nitric oxide; Renal hemodynamics
MeSH Terms: conditions — Heart Failure | interventions — omega-N-Methylarginine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Ng-monomethyl-L-arginine (drug)

SUMMARY:
The study tests the hypothesis that nitric oxide availability is changed in congestive heart failure with regard to the regulation of renal hemodynamics, renal sodium excretion and release of vasoactive hormones. The study tests these hypotheses by comparing the effects of systemic nitric oxide inhibition with L-NMMA in congestive heart failure patients with healthy subjects on renal hemodynamics, blood pressure and plasma levels of vasoactive hormones.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effects of systemic treatment with Ng-monomethyl-l-arginine in congestive heart failure and healthy controls on:

* glomerular filtration rate and renal plasma flow
* blood pressure and heart rate
* plasma levels of vasoactive hormones
* lithium clearance

The study is randomized and placebo controlled

ELIGIBILITY:
Inclusion Criteria:

Healthy controls

* Age 20 to 60 years
* Both men and women
* Weight below 100 kg
* Normal clinical examination and laboratory screening
* Fertile women only if using contraception
* Informed consent according to the regulations of the local ethics committee

Heart failure

* Both men and women
* Age 20 to 75 years
* Patients with heart failure in NYHA group II-III. Heart failure must be derived from ischaemic heart disease or dilated cardiomyopathy. Diagnosis must be verified by history and echocardiography or isotope cardiography.
* ejection fraction < 0.40
* P-creatinin < 250 µmol/L
* Fertile women only if using contraception
* Informed consent according to the regulations of the local ethics committee

Exclusion Criteria:

Healthy controls

* History or clinical evidence of diseases of the heart and blood vessels, kidneys, liver and pancreas, endocrine organs, lungs, neoplastic disease, myocardial infarction or cerebrovascular insult as evaluated by clinical examination and laboratory screening
* Current medication
* Drugs or alcohol abuse
* Pregnancy
* Previously within one year received more than 0.2 mSV radioactive treatment or diagnostic substances
* Donation of blood less than 1 month before the experiments

Heart failure

* Cardiac valvular disease with stenosis
* Significant cardiac arrythmia
* Myocardial infarction, PTCA or by-pass surgery less than 3 months before the study
* Diseases of the lever, kidneys, lungs or endocrine organs which are not secondary to congestive heart failure
* Arterial hypertension
* Neoplastic disease
* Cerebrovascular insult
* Treatment with ACE-inhibitors or nitrates which cannot be stopped 1 week before study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Overall Officials: Jesper N Bech, MD, Ph.D., Principal Investigator — Dept. of Medicine, Holstebro Hospital, 7500 Holstebro, Denmark; Erling B Pedersen, Professor, Study Chair — Dept. of Medicine, Holstebro Hospital, 7500 Holstebro, Denmark